CLINICAL TRIAL: NCT05990920
Title: A Phase 1, Open-Label, Dose Escalation Study of Allogeneic Blood-derived Natural Killer Cells to Evaluate Safety and Tolerability in Participants with Pathologically Confirmed Cancer Refractory to Conventional Therapy
Brief Title: Study of Allogeneic Blood-derived Natural Killer Cells to Evaluate Safety and Tolerability in Cancer Refractory to Conventional Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NKGen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNK02-202
Record Dates: First submitted 2023-07-28; First posted 2023-08-14 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Pathologically Confirmed Cancer Refractory to Conventional Therapy; Refractory Cancer; Metastatic Cancer; Recurrent Cancer; Solid Tumor, Adult; Solid Tumor; Advanced Cancer; Advanced Solid Tumor
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cohort 1 (Experimental): SNK02 will be administered as an IV infusion weekly for 8 weeks.
  Interventions: Biological: SNK02

INTERVENTIONS:
Biological: SNK02 — SNK02 is ex vivo expanded allogeneic NK cells for IV injection, is a light-yellow cryopreserved cell suspension consisting of NK cells isolated from healthy donor's peripheral blood mononuclear cells.

SUMMARY:
The goal of this clinical trial is to test SNK02 in participants with pathologically confirmed cancer that is refractory to conventional therapy. The main questions it aims to answer are:

* Is SNK02 safety and tolerable when administered weekly as an intravenous infusion
* What is the maximum dose that is tolerated of SNK02 Participants will be administered SNK02 weekly for 8 weeks and undergo medical evaluation to provide initial clinical safety data for the treatment of cancer with allogeneic NK cells as a monotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of refractory cancer that has failed at least prior line of conventional standard of care therapy.
* Diagnosed with any histologically confirmed malignancy whose disease is confirmed to be metastatic and/or unresectable for which standard curative or beneficial treatments are no longer effective.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* ≥ 4 weeks since any prior systemic therapy (excluding corticosteroid therapy) to treat the underlying malignancy (standard or investigational).
* ≥ 2 weeks since prior palliative radiotherapy.
* Complete recovery to baseline or Grade 1 NCI CTCAE v5.0 from AE of prior surgery, radiotherapy, endocrine therapy, and other therapy as applicable, with exception of grade 2 alopecia from prior chemotherapy.
* Adequate bone marrow function:

  * Neutrophils: ≥ 1.5 K/µL without colony-stimulating factor support
  * Platelet Count: ≥ 100 K/µL
  * Hemoglobin: ≥ 9.0 g/dL without need for hematopoietic growth factor or transfusion support
  * No ongoing transfusion requirements
* Adequate hepatic function:

  * Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN), does not apply to patients with Gilbert's syndrome
  * Serum albumin ≥ 3.0 g/dL
  * ALT and AST ≤ 2.5 × ULN, unless hepatic metastases are present then < 5 x ULN
* Adequate renal function with creatinine ≤ 2.0 mg/dL.
* Coagulation: INR or aPTT ≤1.5 X ULN unless the subject is receiving anticoagulant therapy.
* Adequate pulmonary function as assessed by pulse oximetry (>92% oxygen saturation on room air).
* Negative pregnancy test for women of childbearing potential (i.e., all women except those who are post menopause for ≥ 1 year or who have a history of hysterectomy or surgical sterilization) and agree to use of effective contraception (hormonal or barrier method of birth control) during study.
* Male participants and female participants of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception

Exclusion Criteria:

* Pregnant and/or lactating females.
* Life expectancy of less than three months.
* Currently being treated by "biological therapy" as defined by the National Cancer Institute (https://www.cancer.gov/about-cancer/treatment/types/immunotherapy/bio-therapies-fact-sheet) Examples include checkpoint inhibitors, adoptive cell transfer, monoclonal antibodies, treatment vaccines, cytokines, CAR-T therapy, and natural killer (NK) cell therapy.
* Participants that are actively positive for COVID.
* Autoimmune disease requiring therapy; immunodeficiency, or any disease process requiring immunosuppressive therapy, with exception to the following:

  * intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection);
  * Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent;
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* Prior clinical trial requiring participant to receive an investigational drug within four weeks of enrollment.
* Live vaccine within 30 days prior to enrollment.
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* Mental or psychological illness preventing cooperation with treatment, efficacy evaluations.
* Participants who have undergone prior organ transplantation, including allogeneic stem-cell transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicity as assessed by labs, PE and AEs | 4 weeks
  Evaluate the safety and tolerability of SNK02 assessed by labs, PE and AEs
MTD and/or RP2D | 8 weeks
  Determine the maximum tolerated dose or the ready for Phase 2 dose of SNK02
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 12 weeks
  Evaluate the safety and tolerability of SNK02 assessed by labs, PE and AEs

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Angeles Clinic and Research Institute, Los Angeles, California
  - Sarcoma Oncology Center, Santa Monica, California

IPD SHARING:
Plan to Share IPD: No